CLINICAL TRIAL: NCT03083600
Title: A Randomized, Double-blind, Placebo-controlled, Study to Assess Efficacy and Safety of Protein Hydrolysates in the Reduction and Maintenance of HbA1c Levels in a Pre-diabetic Population
Brief Title: Effect of Protein Hydrolysates on HbA1c Levels in Pre-diabetics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Study was not recruiting
Sponsor: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFCRO-071
Record Dates: First submitted 2017-02-27; First posted 2017-03-20 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: PreDiabetes
Keywords: protein hydrolysates; HbA1c; prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: 56 participants randomised to receive: 5g, 10g, 15g Pea Protein Hydrolysate v placebo 5g, 10g, 15g v Rice Protein Hydrolysate v placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, computer-generated randomisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Plant-based Protein Hydrolysate (1) 5g (Active Comparator): plant-based protein hydrolysate 1 (5g) stored in aluminium sachets to be reconstituted with 100 mL of water and administered 2 times per day for 12-weeks
  Interventions: Dietary Supplement: Plant-based Protein Hydrolysate 1
- Plant-based Protein Hydrolysate (1) 10g (Active Comparator): Plant-based protein hydrolysate 1 (10 g) stored in aluminium sachets to be reconstituted with 100 mL of water and administered 2 times daily for 12-weeks
  Interventions: Dietary Supplement: Plant-based Protein Hydrolysate 1
- Plant-based Protein Hydrolysate (1) 15 g (Active Comparator): Plant-based 1 protein hydrolysate (15 g) stored in aluminium sachets to be reconstituted with 100 mL of water and administered 2 times daily for 12-weeks
  Interventions: Dietary Supplement: Plant-based Protein Hydrolysate 1
- Placebo (Placebo Comparator): Cellulose Placebo stored in aluminium sachets to be reconstituted with 100 mL of water and administered 2 times daily for 12-weeks.
  Interventions: Dietary Supplement: Placebo
- Plant-based Protein Hydrolysate (2) 5g (Active Comparator): Plant-based protein hydrolysate 2 (5 g) stored in aluminium sachets to be reconstituted with 100 mL of water and administered 2 times daily for 12-weeks
  Interventions: Dietary Supplement: Plant-based Protein Hydrolysate 2
- Plant-based Protein Hydrolysate (2) 10g (Active Comparator): Plant-based protein hydrolysate 2 (10 g) stored in aluminium sachets to be reconstituted with 100 mL of water and administered 2 times daily for 12-weeks
  Interventions: Dietary Supplement: Plant-based Protein Hydrolysate 2
- Plant-based Protein Hydrolysate (2) 15g (Active Comparator): Plant-based protein hydrolysate 2 (15 g) stored in aluminium sachets to be reconstituted with 100 mL of water and administered 2 times daily for 12-weeks
  Interventions: Dietary Supplement: Plant-based Protein Hydrolysate 2

INTERVENTIONS:
Dietary Supplement: Plant-based Protein Hydrolysate 1 — Plant-based Protein Hydrolysate 2 for 12-weeks
  Arms: Plant-based Protein Hydrolysate (1) 10g; Plant-based Protein Hydrolysate (1) 15 g; Plant-based Protein Hydrolysate (1) 5g
Dietary Supplement: Plant-based Protein Hydrolysate 2 — Plant-based Protein Hydrolysate 2 for 12-weeks
  Arms: Plant-based Protein Hydrolysate (2) 10g; Plant-based Protein Hydrolysate (2) 15g; Plant-based Protein Hydrolysate (2) 5g
Dietary Supplement: Placebo — Cellulose Placebo for 12-weeks
  Arms: Placebo

SUMMARY:
To evaluate the effectiveness of three different daily doses of plant protein hydrolysates versus placebo, when consumed over a 12-week period, at reducing and maintaining glycated haemoglobin (HbA1c) levels in a pre-diabetic population (otherwise healthy subjects with impaired glucose metabolism).

To evaluate the effectiveness of three different daily doses of pea or rice protein hydrolysates versus placebo, when consumed over a 12-week period on: post-prandial glucose/insulin levels (oral glucose tolerance test, fructosamine levels, fasting plasma glucose levels, vital signs, physical examinations, weight and blood pressure.

DETAILED DESCRIPTION:
Diabetes has been recognised as an epidemic globally and within the EU. Environmental and behavioural changes over the last century, such as a sedentary lifestyle, intake of calorie dense/sugary foods and obesity are all significant contributors in creating a dramatic increase in the incidence of diabetes globally. There are about 60 million people, 11% of the total population, with diabetes in the European Region. This number will swell to 15% of the EU population by 2030. Europe spent €89 billion on directly treating and managing diabetes and its related complications in 2011. This cost however is severely understated as the true cost of diabetes also includes indirect costs, such as productivity losses due to lost working time through absenteeism, sickness, early retirement and premature death. The WHO projects that diabetes will be the 7th leading cause of death in 2030 and it is already the fourth in most developed countries in the world.

Additionally, individuals with diabetes are twice as likely to be admitted to hospital. According to the International Diabetes Federation (IDF), diabetes is the number one cause for admission to dialysis and to kidney transplant programmes and is the leading cause of working age blindness. It also accounts for a risk of lower limb amputation of 10 to 12%. Therefore, it is clear that diabetes has a huge and growing impact on individual sufferers as well as placing a huge strain on the health system and the exchequers that have to fund them.

90% of diabetes patients globally have type 2 diabetes and when we refer to diabetes in the document going forward it is type 2 to which we refer. This chronic disease state occurs when the body does not use insulin properly causing glucose levels in the blood to rise higher than normal. This abnormal state over time leads to serious damage to the heart, blood vessels, eyes, kidneys, and nerves. Prediabetic individuals are defined as having blood sugar levels higher than normal but not yet high enough to be classified as Diabetes, and prediabetes is thought of as a clear, early warning sign for diabetes.

Without intervention, prediabetes is likely to become type 2 diabetes in 10 years or less. The increasing number of new cases of prediabetes presents a global concern as it carries large-scale implications towards the future burden on healthcare. Between 2003 and 2011, the prevalence of prediabetes in England alone more than tripled, with 35.3% of the adult population, or 1 in every 3 people, having prediabetes. The International Journal of health science succinctly states a well-accepted fact: "intervention prior to the onset of type 2 diabetes may be the only way of preventing the complications of diabetes". In addition, diabetes once it occurs is irreversible, thus prevention holds a last beacon for epidemic control in the future.

Whilst significant lifestyle changes can be impactful, sustained compliance is very limited and therefore results are poor. As a result, the European Commission has highlighted functional foods as valuable solutions for treatment and prevention of diabetes. A functional food, "beneficially affects one or more target functions in the body beyond adequate nutritional effects in a way that is relevant to either an improved state of health and well-being and/or reduction of risk of disease.

Peptides derived from a range of food materials have been shown to prevent disease i.e. inflammatory disorders [1] osteoporosis [2] high blood pressure [3] or promote health i.e. immunomodulatory [4], antimicrobial [5], anti-oxidative [6], antithrombotic [7], hypo-cholesterolemic [8] activities.

Peptides are protein molecules smaller than 10 kDa that may exist naturally or be derived from full length proteins. Bioactive peptides are defined as specific protein fragments that have positive effects on body functions or conditions and may influence human health [9]. Peptides are produced by hydrolysis of food materials by digestive, microbial, and plant proteolytic enzymes, their levels generally increase during food fermentation [10]. Bioactive peptides with particular amino-acid sequences, which are inactive in the intact protein molecule become bioactive after their release from the intact molecule through the action of digestive enzymes in the body or through the action of proteolytic enzymes in food processing.

Plant hydrolysates have been shown to display a stimulatory effect on the insulin responsive glucose transport protein, GLUT4, which facilitates glucose transport into skeletal muscle. Skeletal muscle is the predominant site of glucose disposal (80%) under insulin-stimulated or post-prandial conditions and so it is hypothesized that one or both of the Nuritas pea and rice protein hydrolysates could help reduce HbA1c levels in those with elevated HbA1c levels (prediabetes).

The main aims are to evaluate the effectiveness of three different daily doses of plant-based hydrolysates versus placebo, when consumed over a 12-week period, at reducing and maintaining glycated haemoglobin (HbA1c) levels in a pre-diabetic population (otherwise healthy subjects with impaired glucose metabolism), as well as post-prandial glucose/insulin levels (oral glucose tolerance test), fructosamine levels, fasting plasma glucose levels, vital signs, physical examinations, weight, blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent,
2. Be aged between 18 and 75 years, inclusive,
3. Have a HbA1c of > 5.7% and < 6.4% (38.8mmol/L - 47mmol/L),
4. Be a non-smoker,
5. Have a body mass index (BMI) 20 - 35 kg/m²,
6. Have a stable bodyweight (+/- 5%) in the last 3 months,
7. Not currently taking regular supplements (within 1 month of study entry),
8. Be willing to maintain dietary habits and physical activity levels throughout the trial period,
9. Be able to communicate well with the Investigator, to understand and comply with the requirements of the study, and be judged suitable for the study in the opinion of the Investigator.

Exclusion Criteria:

1. Diagnosed diabetes with a HbA1c >6.4% (47mmol/l)
2. Body Mass Index (BMI) less than 20 (underweight) or greater than 35 (morbidly obese)
3. Have a significant acute or chronic coexisting illness such as cardiovascular disease, chronic kidney or liver disease, gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease or any condition which contraindicates, in the investigators judgement, entry to the study
4. Consumption of more than the recommended alcohol guidelines i.e. >21 alcohol units/week for males and >14 units/week for females
5. Currently or recently (within 3 months of study entry) taking any medication, which in the opinion of the investigator, could interfere with the outcome of the study, including insulin and acetylsalicylic acid
6. If subjects are taking hypolipidemic agents and/or beta-blockers, their dose must be stable for greater than 3 months,
7. Known allergy to any of the components of the test product
8. History of drug or alcohol abuse
9. Present or recent use (within 3 months of screening) of dietary supplements that affect the level of blood glucose, e.g chromium,
10. Low hemoglobin or hematocrit (i.e., lower than accepted laboratory values),
11. Females are pregnant, lactating or wish to become pregnant during the study. Female subject is currently either of:

    * non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or any female who is surgically sterilized (via documented hysterectomy or bilateral tubal ligation). (For purposes of this study, postmenopausal is defined as one year without menses), OR
    * child bearing potential, the subject is eligible to enter and participate in this study if she is not lactating and has a negative urine pregnancy test at the screening visit, visit 2 and upon completion of the study at visit 5. The subject must also agree to one of the following methods of contraception: i. Complete abstinence from intercourse two weeks prior to administration of study drug, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study medication in cases where subject discontinues the study prematurely. (Subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit.) or, ii. has a male sexual partner who is surgically sterilized prior to the Screen Visit and is the only male sexual partner for that subject or, iii. sexual partner(s) is/are exclusively female or, iv. Oral contraceptives (either combined or progestogen only) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm. (Women of child-bearing potential using an oral contraceptive in combination with a double-barrier method of contraception are required to continue to use this form of contraception for 1 week following discontinuation of study medication).

      v. Use of double-barrier contraception, specifically, a spermicide plus a mechanical barrier (e.g. male condom, female diaphragm). The subject must be using this method for at least 1 week following the end of the study or, vi. Use of any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year. The subject must have the device inserted at least 2 weeks prior to the first Screen Visit, throughout the study, and 2 weeks following the end of the study.
12. Participation in a clinical trial with an investigational product within 90 days before screening, or plans to participate in another study during the study period,
13. Subject has a history of non-compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Plasma Glycated Haemoglobin (HbA1c) (mmol/mol) | 12-weeks
  5, 10, 15 g Plant-based protein hydrolysate (1 or 2) vs placebo

SECONDARY OUTCOMES:
Post-prandial blood glucose (mmol/L) | 12-weeks
  5, 10, 15 g pea and rice protein hydrolysate vs placebo
Post-prandial blood insulin (pmol/L) | 12-weeks
  5, 10, 15 g Plant-based protein hydrolysate (1 or 2) vs placebo
Weight (kg) | 12-weeks
  5, 10, 15 g Plant-based protein hydrolysate (1 or 2) vs placebo
Blood pressure (mmHg) | 12-weeks
  5, 10, 15 g Plant-based protein hydrolysate (1 or 2) vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Shanahan, MD, Principal Investigator — Cork University Hospital
Locations (1):
- Atlantia Food Clinical Trials, University College Cork, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No